CLINICAL TRIAL: NCT06232837
Title: Macintosh Blade Size During Laryngoscopy for Endotracheal Intubation in Operative Rooms. A Nationwide Prospective Observational Study.
Brief Title: Macintosh Blade Size for Endotracheal Intubation in Operative Rooms
Acronym: MacSize_OR
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Société Française d'Anesthésie-Réanimation (SFAR) (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB 00010254-2023-081
Record Dates: First submitted 2024-01-10; First posted 2024-01-31 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-11

CONDITIONS: Intubation Complication; Intubation; Difficult or Failed; Endotracheal Intubation
Keywords: Intubation; Operative Room; Macintosh; Direct Laryngoscopy; Video Laryngoscopy; Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Macintosh blade size 3: Patients intubated using Macintosh blade size 3
  Interventions: Device: Direct laryngoscopy using Macintosh blade
- Macintosh blade size 4: Patients intubated using Macintosh blade size 4
  Interventions: Device: Direct laryngoscopy using Macintosh blade

INTERVENTIONS:
Device: Direct laryngoscopy using Macintosh blade — Patients in operative room requiring direct laryngoscopy for endotracheal intubation

SUMMARY:
Endotracheal intubation is a frequent procedure in the operating room but optimal Macintosh blade size remains unknown to date.

DETAILED DESCRIPTION:
Endotracheal intubation is an extremely frequent procedure in the operating room, in intensive care units and in emergency medicine (in- or out-of-hospital). Apart from special cases of foreseen difficult programmed intubation, direct laryngoscopy remains the most frequently used technique. It requires the use of a handle (short or long), which serves as a light source on which is adapted a Macintosh curved blade, metallic or plastic, single or multiple use. The choice of blade size is based on the experience of the physician. Most often, in adult settings, size 3 or 4 blades are used. The very spartan literature on the subject and the current recommendations do not provide any information on the choice of blade size. Our team (and others) recently concluded that intubation first attempt rates in intensive care units or emergency settings were improved when using shorter Macintosh blade size No3 vs 4 (Godet et al. Intensive Care Medicine 2022 and Landefeld et al. Critical Care Explorations 2023). We therefore wish to evaluate these practices in terms of success of the first laryngoscopy, Cormack-Lehane and POGO (percentage of glottic opening visualized) scores, the need to use an alternative technique or a second operator in operative rooms. The results will be analyzed with regard as a function and experience of the person performing the laryngoscopy, as well as the setting (urgent or scheduled). These data are usually collected during the performance of an endotracheal intubation in a nationwide fashion in French operative rooms.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be admitted in a participating operative room and require mechanical ventilation through an orotracheal tube.
* Adult (age ≥ 18 years)
* Subjects must be covered by public health insurance
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Anticipated difficult intubation requiring videolaryngoscopy or other technic in first place
* Nasotracheal intubation
* Refusal of study participation or to pursue the study by the patient
* Absence of coverage by the French statutory healthcare insurance system
* Protected person

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any patient requiring orotracheal intubation with direct laryngoscopy in first place
Sampling Method: Non-Probability Sample
Enrollment: 3058 (Actual)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-09-20 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Number of patients with successful first-pass orotracheal intubation | At intubation
  The proportion of patients with successful first-pass orotracheal intubation

SECONDARY OUTCOMES:
Severe complications related to intubation_hypoxemia | At intubation
  Rate of severe hypoxemia defined by lowest oxygen saturation (SpO2) < 90 %
Severe complications related to intubation_severe collapse | At intubation
  Rate of cardiovascular collapse, defined as systolic blood pressure less than 80 mmHg systolic blood pressure less than 50 mmHg recorded at least once
Severe complications related to intubation_cardiac arrest | At intubation
  Rate of cardiac arrest related to intubation
Severe complications related to intubation_death | At intubation
  Rate of death related to intubation
Moderate complications related to intubation_difficult intubation | At intubation
  Rate of difficult intubation
Moderate complications related to intubation_arrythmia | At intubation
  Rate of severe ventricular or supraventricular arrhythmia requiring intervention
Moderate complications related to intubation_oesophageal intubation | At intubation
  Rate of oesophageal intubation
Moderate complications related to intubation_agitation | At intubation
  Rate of agitation
Moderate complications related to intubation_aspiration | At intubation
  Rate of pulmonary aspiration
Moderate complications related to intubation_dental injuries | At intubation
  Rate of dental injuries
Cormack Lehane | During laryngoscopy
  Cormack-Lehane grade of glottic view
Percentage of Glottic Opening | During laryngoscopy
  Percentage of Glottic Opening (POGO) grade of glottic view
Difficulty of intubation | During intubation
  Rate of operator-assessed difficulty of intubation
Additional airway equipment | During intubation
  Rate of need for additional airway equipment (video laryngoscope, bougie, stylet, fibroscope, cricothyrotomy)
Additional second operator | During intubation
  Rate of need for a second operator

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Godet, MD, PhD, Principal Investigator — Clermont-Ferrand University Hospitals
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: Yes
Data available upon reasonable request and satisfactory presented analysis plan. Authorship will include principal investigator (last author).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data available after study completion and publication

REFERENCES:
- [Background] Godet T, De Jong A, Garin C, Guerin R, Rieu B, Borao L, Pereira B, Molinari N, Bazin JE, Jabaudon M, Chanques G, Futier E, Jaber S. Impact of Macintosh blade size on endotracheal intubation success in intensive care units: a retrospective multicenter observational MacSize-ICU study. Intensive Care Med. 2022 Sep;48(9):1176-1184. doi: 10.1007/s00134-022-06832-9. Epub 2022 Aug 16. PMID 35974189
- [Background] Landefeld KR, Koike S, Ran R, Semler MW, Barnes C, Stempek SB, Janz DR, Rice TW, Russell DW, Self WH, Vonderhaar D, West JR, Casey JD, Khan A. Effect of Laryngoscope Blade Size on First Pass Success of Tracheal Intubation in Critically Ill Adults. Crit Care Explor. 2023 Mar 6;5(3):e0855. doi: 10.1097/CCE.0000000000000855. eCollection 2023 Mar. PMID 36895888